CLINICAL TRIAL: NCT03841890
Title: The Clarus Video System (Trachway) and Direct Laryngoscope for Endotracheal Intubation With Cricoid Pressure in Simulated Rapid Sequence Induction Intubation: A Prospective Randomized Controlled Trial
Brief Title: The Clarus Video System and Direct Laryngoscope for Rapid Sequence Induction Intubation With Cricoid Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201601025A3C502
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2016-11

CONDITIONS: Intubation, Intratracheal; Laryngoscopes; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sore throat and mucosa injury are documented by a blinded observer on the next day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intubation with the Clarus Video System as a video stylet (Experimental)
  Interventions: Device: the Clarus Video System as a video stylet
- Intubation with the Clarus Video System as a lightwand (Experimental)
  Interventions: Device: the Clarus Video System as a lightwand
- Intubation with direct laryngoscope (Active Comparator)
  Interventions: Device: direct laryngoscope

INTERVENTIONS:
Device: the Clarus Video System as a video stylet — video-guided intubation
  Other Names: Trachway as a video stylet
  Arms: Intubation with the Clarus Video System as a video stylet
Device: the Clarus Video System as a lightwand — The endotracheal tube will be initially guided into larynx in the dimly lit operating room by a bright glow moving in the anterior soft tissue of the neck and finally by the image of the trachea rings on the video screen.
  Other Names: Trachway as a lightwand
  Arms: Intubation with the Clarus Video System as a lightwand
Device: direct laryngoscope — Macintosh laryngoscope size 3
  Arms: Intubation with direct laryngoscope

SUMMARY:
During an emergency endotracheal intubation, rapid sequence induction intubation with cricoid pressure is frequently implemented to prevent aspiration pneumonia. When properly applied, cricoid pressure may not affect glottic view during endotracheal intubation with either a direct laryngoscope or a video laryngoscope. However, the application of cricoid pressure is likely to prolong the intubation time. Limited mouth opening or vulnerable teeth, which often accompany the patients requiring emergency intubation, are the two common factors to deter the intubators from using a laryngoscopic device. Besides, the blade of a laryngoscopic device is often too bulky for a narrow mouth opening, and the blade always bears a level force on upper incisors while the intubator is lifting epiglottis during intubation, which is liable to tooth fracture. In this prospective randomized study, the investigators compare the use of the Clarus Video System and that of direct laryngoscope (Macintosh Laryngoscope) in patients undergoing endotracheal intubation in simulated rapid sequence induction intubation for the primary goals of the first attempt success rate and intubation time.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years of age
* Scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* BMI (Body Mass Index) > 35 kg/m2
* Interincisor distance < 3 cm
* Poor dentition
* Upper airway tumor
* Limited neck mobility
* Pregnancy
* History of difficult tracheal intubation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-14 (Actual)

PRIMARY OUTCOMES:
The first attempt success rate | After intubation immediately
Intubation time | After intubation immediately
  Intubation time was counted from the inserting the device into the patient's mouth to viewing the endotracheal tube into the trachea.

SECONDARY OUTCOMES:
Blood pressure | 1 minute and 5 minutes after intubation
  Measure blood pressure in millimeter of mercury by non-invasive blood pressure before induction, 1 minute after intubation, and 5 minutes after intubation
Heart rate | 1 minute and 5 minutes after intubation
  Measure heart rate in beats per minute by electrocardiography monitor before induction, 1 minute after intubation, and 5 minutes after intubation
Sore throat | On postoperative day 1
  Documented by a blinded observer on the next day. Sore throat was graded according to numerical rating scale (NRS): none, NRS = 0; mild, NRS = 1-3; moderate, NRS = 4-6; severe, NRS = 7-10.
Mucosal injury | On postoperative day 1
  Documented by a blinded observer on the next day. "Yes" is defined as any oral mucosal lesion reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: An-Hsun Cho, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Algie CM, Mahar RK, Tan HB, Wilson G, Mahar PD, Wasiak J. Effectiveness and risks of cricoid pressure during rapid sequence induction for endotracheal intubation. Cochrane Database Syst Rev. 2015 Nov 18;2015(11):CD011656. doi: 10.1002/14651858.CD011656.pub2. PMID 26578526
- [Background] Birenbaum A, Hajage D, Roche S, Ntouba A, Eurin M, Cuvillon P, Rohn A, Compere V, Benhamou D, Biais M, Menut R, Benachi S, Lenfant F, Riou B; IRIS Investigators Group. Effect of Cricoid Pressure Compared With a Sham Procedure in the Rapid Sequence Induction of Anesthesia: The IRIS Randomized Clinical Trial. JAMA Surg. 2019 Jan 1;154(1):9-17. doi: 10.1001/jamasurg.2018.3577. PMID 30347104
- [Background] Sajayan A, Wicker J, Ungureanu N, Mendonca C, Kimani PK. Current practice of rapid sequence induction of anaesthesia in the UK - a national survey. Br J Anaesth. 2016 Sep;117 Suppl 1:i69-i74. doi: 10.1093/bja/aew017. Epub 2016 Feb 24. PMID 26917599
- [Background] Vanner RG, Clarke P, Moore WJ, Raftery S. The effect of cricoid pressure and neck support on the view at laryngoscopy. Anaesthesia. 1997 Sep;52(9):896-900. doi: 10.1111/j.1365-2044.1997.181-az0315.x. PMID 9349075
- [Background] Turgeon AF, Nicole PC, Trepanier CA, Marcoux S, Lessard MR. Cricoid pressure does not increase the rate of failed intubation by direct laryngoscopy in adults. Anesthesiology. 2005 Feb;102(2):315-9. doi: 10.1097/00000542-200502000-00012. PMID 15681945
- [Background] Komasawa N, Kido H, Miyazaki Y, Tatsumi S, Minami T. Cricoid pressure impedes tracheal intubation with the Pentax-AWS Airwayscope(R): a prospective randomized trial. Br J Anaesth. 2016 Mar;116(3):413-6. doi: 10.1093/bja/aev438. Epub 2016 Jan 27. PMID 26821697
- [Background] Byhahn C, Nemetz S, Breitkreutz R, Zwissler B, Kaufmann M, Meininger D. Brief report: tracheal intubation using the Bonfils intubation fibrescope or direct laryngoscopy for patients with a simulated difficult airway. Can J Anaesth. 2008 Apr;55(4):232-7. doi: 10.1007/BF03021507. PMID 18378968
- [Background] Hung OR, Pytka S, Morris I, Murphy M, Launcelott G, Stevens S, MacKay W, Stewart RD. Clinical trial of a new lightwand device (Trachlight) to intubate the trachea. Anesthesiology. 1995 Sep;83(3):509-14. doi: 10.1097/00000542-199509000-00009. PMID 7661351
- [Background] Cooney DR, Beaudette C, Clemency BM, Tanski C, Wojcik S. Endotracheal intubation with a video-assisted semi-rigid fiberoptic stylet by prehospital providers. Int J Emerg Med. 2014 Nov 26;7(1):45. doi: 10.1186/s12245-014-0045-0. eCollection 2014. PMID 25593618
- [Background] Yang M, Kim JA, Ahn HJ, Choi JW, Kim DK, Cho EA. Double-lumen tube tracheal intubation using a rigid video-stylet: a randomized controlled comparison with the Macintosh laryngoscope. Br J Anaesth. 2013 Dec;111(6):990-5. doi: 10.1093/bja/aet281. Epub 2013 Aug 23. PMID 23975566
- [Background] Hsu HT, Chou SH, Chen CL, Tseng KY, Kuo YW, Chen MK, Cheng KI. Left endobronchial intubation with a double-lumen tube using direct laryngoscopy or the Trachway(R) video stylet. Anaesthesia. 2013 Aug;68(8):851-5. doi: 10.1111/anae.12340. PMID 24044439
- [Background] Hodgson RE, Gopalan PD, Burrows RC, Zuma K. Effect of cricoid pressure on the success of endotracheal intubation with a lightwand. Anesthesiology. 2001 Feb;94(2):259-62. doi: 10.1097/00000542-200102000-00015. PMID 11176090
- [Derived] Lin YC, Cho AH, Lin JR, Chung YT. The Clarus Video System (Trachway) and direct laryngoscope for endotracheal intubation with cricoid pressure in simulated rapid sequence induction intubation: a prospective randomized controlled trial. BMC Anesthesiol. 2019 Mar 4;19(1):33. doi: 10.1186/s12871-019-0703-0. PMID 30832590